CLINICAL TRIAL: NCT00484601
Title: Phase II Study of Ifosfamide and Doxorubicin in Patients With Refractory Nasopharyngeal Carcinoma
Brief Title: Ifosfamide and Doxorubicin in Patients With Refractory Nasopharyngeal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS0327; 03-09-11-08 (Other: JHM IRB)
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Refractory Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Ifosfamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ifosfamide and Doxorubicin (Experimental): Single arm treatment with Ifosfamide and Doxorubicinin patients with Refractory Nasopharyngeal Carcinoma
  Interventions: Drug: Ifosfamide; Drug: Doxorubicin

INTERVENTIONS:
Drug: Ifosfamide
Drug: Doxorubicin

SUMMARY:
This research is to test the effectiveness and toxicity of both Ifosfamide and Doxorubicin. It also aims to explore the relationship between EBV DNA and clinical response in patients with advanced naso-pharyngeal cancer which has been previously treated with chemotherapy.

DETAILED DESCRIPTION:
Nasopharyngeal Cancer (NPC) is one of the common cancer in Southeast Asia. In this region NPC is associated with Epstein Barr Virus (EBV) chronic infection with EBV DNA identifiable in almost all the NPC tumors and patient's serum at the time of diagnosis. Chinese, especially cantonese has the highest incidence. Only about 30% of patients presents early disease and has a good treatment outcome (80% cure for stage I disease and 70% for stage II by radiation).

This research is to test the effectiveness and toxicity of both Ifosfamide and Doxorubicin. It also aims to explore the relationship between EBV DNA and clinical response in patients with advanced naso-pharyngeal cancer which has been previously treated with chemotherapy.

Investigators believe EBV infection is necessary to cause NPC and that EBV DNA levels in the blood may directly relate to the total size of the tumor. Because NPC patients in this situation have a poor outlook, we design this study to evaluate the combination of Ifosfamide and doxorubicin for further treatment. While this combination of medicines has been used in many other forms of cancer, it has not been tested in patients with NPC.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of NPC
* Age > 18 years old
* Measurable metastatic or recurrent disease (s)
* Received one prior chemotherapy regimen for metastatic or recurrent NPC which relapsed or became refractory before entry.
* ECOG PS 0, 1 or 2
* WBC > 3,500/uL and ANC > 1,500/uL Platelet > 100,000/uL Creatinine - within normal limits SGOT < 3 X UNL Bilirubin < 2.0 mg/dL
* Ejection fraction > 45% and no history of myocardial infarction or congestive heart failure in the last 6 months. No history of cardiac ventricular arrythmia or ventricle tachycardia, or uncontrolled atrial fibrillation or supraventricular tachycardia with hemodynamic compromising status.
* Random blood glucose level < 250 mg
* Signed informed consent

Exclusion Criteria:

* Received more than one prior chemotherapy for metastatic or recurrent disease
* Ejection fraction < 45%
* WBC < 3,500/UL or ANC < 1,500/UL or P/t < 100,000/UL or SCOT> 3 x UNL or Bilirubin > 2.0 mg/dL or Creatinine > UNL
* ECOG PS > 3
* Hx of myocardial infarction within last 6 months
* Random blood glucose level less than or equal 250 mg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-04-15 (Actual); Primary Completion 2007-11-07 (Actual); Study Completion 2007-11-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall response rate and toxicity including complete response rate, response duration, time to treatment failure, and survival of ifosfamide and doxorubicin as the second line chemotherapy for patients with advanced NPC | May 2008
  Prematured termination, data is not analysed.

SECONDARY OUTCOMES:
To correlate EBVDNA titer with clinical response | May 2008
  Prematured termination, data is not analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chang, MD, Principal Investigator — Johns Hopkins Singapore
Locations (1):
- Johns Hopkins Singapore International Medical Center, Singapore, Singapore